CLINICAL TRIAL: NCT07173530
Title: Low Level Light Therapy & Skin Pigmentation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Eric R. Ritchey, Associate Professor, University of Houston
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005386/MOD00007330
Record Dates: First submitted 2025-07-07; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-07

CONDITIONS: Dry Eye; Meibomian Gland Dysfunction (Disorder)
Keywords: Dry Eye; Meibomian Gland; LLLT; Low-level light therapy
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Fitzpatrick skin tone I-IV (Experimental): Individuals with skin tones I-IV on the Fitzpatrick scale will receive low-level light therapy
  Interventions: Device: Three 15-minute low-level light therapy sessions using Light Emitting Diodes of wavelength 633nm (Essilor epi-c plus).
- Fitzpatrick skin tone V-VI (Experimental): Individuals with skin tones V-Vi on the Fitzpatrick scale will receive low-level light therapy
  Interventions: Device: Three 15-minute low-level light therapy sessions using Light Emitting Diodes of wavelength 633nm (Essilor epi-c plus).

INTERVENTIONS:
Device: Three 15-minute low-level light therapy sessions using Light Emitting Diodes of wavelength 633nm (Essilor epi-c plus). — A mask with Light Emitting Diodes wavelength 633nm will be placed over closed eyes for 15 minutes.

SUMMARY:
The goal of this clinical trial is to determine if there is a difference in eyelid temperature after low-level light therapy (LLLT) in individuals with different amounts of skin pigmentation and dry eye/meibomian gland disease. Participants will have 3 fifteen minute in office LLLT therapy sessions over a period of approximately 7 to 14 days.

DETAILED DESCRIPTION:
The primary objective of the study is to determine if there is a difference in the thermal effect of low-level light therapy (LLLT) in individuals with different skin pigmentation (Fitzpatrick skin type I-IV verses Fitzpatrick skin type V-VI) using a clinically available 633nm LLLT system, the Epi-C-Plus (Espansione group, Bologna, Italy).

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and understand the study informed consent in English
* Age 18 years or older at enrollment
* Individuals with MGD based on one or more of the following clinical signs/symptoms, e.g., meibum quality score of 1-3 (Bron et al.), meibography score of 1, 2, or 3 on the Pult Meiboscale, non-invasive 1st tear break up time of 10 seconds or less, or an Ocular Surface Disease Index (OSDI) score greater than 12 points.

Exclusion Criteria:

* Active anterior segment pathology (e.g., bacterial conjunctivitis, microbial keratitis)
* History of systemic disease associated with aqueous-deficient dry eye disease (e.g., Sjogren's syndrome)
* History of corneal surgery, refractive surgery, or eyelid surgery within 6 months
* History of corneal ectasia (e.g. keratoconus, Pellucid marginal degeneration)
* History of ocular trauma within 6 months
* History of LipiFlow, iLux, Meiboflow, IPL or LLLT within the last 12 months
* Habitual use of photosensitizing medications within the last 30 days
* Pregnant and/or lactating females, by self-report
* Pigmented lesions, tattoos, or skin cancer in the periocular region
* Unwilling to have eyes photographed or video recorded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Eyelid temperature | Eyelid temperature will be measured before and after 15 minutes of low-level light therapy at the baseline visit.

SECONDARY OUTCOMES:
Ocular Surface Disease Index Questionnaire | After 3 low-level light therapy treatment sessions through study completion, an average of 1 week.
Tear break up time | After 3 low-level light therapy treatment sessions through study completion, an average of 1 week.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Houston College of Optometry, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided